CLINICAL TRIAL: NCT06312384
Title: The Influence of 3D Surgical Template on the Contour of Bone Augmentation, in Patients With Labial Alveolar Ridge Defect and Simultaneous Implantation
Brief Title: The Influence of 3D Surgical Template on the Contour of Bone Augmentation, in Patient With Labial Alveolar Ridge Defect and Simultaneous Implantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A04080622
Record Dates: First submitted 2024-02-29; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-12

CONDITIONS: Bone Deformity
Keywords: 3D surgical template, guided bone regeneration , the contour of bone augmentation ,horizontal labial ridge defect and simultaneous implantation.

STUDY DESIGN:
Intervention Model Description: Group 1 [Control group]:
  The defected site will be grafted with sticky bone (particulate bone substitute mixed with injectable platelet-rich fibrin (i-PRF)) and will be covered with collagen membrane will be applied [conventional GTR].
  Group 2 [Study group]:
  The defected site will be grafted with sticky bone (particulate bone substitute mixed with injectable platelet-rich fibrin (i-PRF)) and will be covered with collagen membrane will be applied, in this group 3D surgical template will be applied.
Who Masked: Outcomes Assessor
Masking Description: each patient will be couded and only the princeiple investigator is the only person how know the type of intervantion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Active Comparator): The defected site will be grafted with sticky bone (particulate bone substitute mixed with injectable platelet-rich fibrin (i-PRF)) and will be covered with collagen membrane will be applied, in this group 3D surgical template will be applied which consist of a two-piece tooth-supported surgical template will fabricated through 3D printing technology before surgery base on the digital simulation of bone graft contour.
  Interventions: Procedure: 3D Surgical Template on the Contour of Bone Augmentation, in Patient With Labial Alveolar Ridge Defect and Simultaneous Implantation
- control (Active Comparator): The defected site will be grafted with sticky bone (particulate bone substitute mixed with injectable platelet-rich fibrin (i-PRF)) and will be covered with collagen membrane will be applied [conventional guided tissue regeneration].
  Interventions: Procedure: conventional guided bone regeneration,in Patient With Labial Alveolar Ridge Defect and Simultaneous Implantation

INTERVENTIONS:
Procedure: 3D Surgical Template on the Contour of Bone Augmentation, in Patient With Labial Alveolar Ridge Defect and Simultaneous Implantation — a two-piece tooth-supported surgical template will fabricated through 3D printing technology before surgery base on the digital simulation of bone graft contour.Sticky bone will placed into the defect under the guidance of the template to form customized sticky bone and will be covered with collagen membrane.
  Arms: study
Procedure: conventional guided bone regeneration,in Patient With Labial Alveolar Ridge Defect and Simultaneous Implantation — The defected site will be grafted with sticky bone (particulate bone substitute mixed with injectable platelet-rich fibrin (i-PRF)) and will be covered with collagen membrane.
  Arms: control

SUMMARY:
Evaluate the impact of using 3D surgical template with guided bone regeneration technique on the contour of bone augmentation in patients with horizontal labial ridge defect and simultaneous implantation.

DETAILED DESCRIPTION:
Because adequate bone wrapping around the implant is critical for long-term effectiveness of dental implant treatment, bone augmentation in the bone defect area is required to repair the width and height of the alveolar bone, as bone resorption occurs following tooth extraction.

Many bone augmentation techniques, such as onlay block grafting, bone splitting, distraction osteogenesis, and guided bone regeneration, are currently accessible in clinics (GBR). Surgical options vary depending on the severity of the bone deformity. GBR is a bone augmentation technique that has more evidence-based medicine support and therapeutic applications, as well as the benefits of less surgical stress and low technical sensitivity.

Establishing aesthetics and guaranteeing long-term success in implant therapy can be challenging. Long-term stable implant success has been linked to the presence of more than 2mm labial graft thickness, and appropriate labial graft thickness is essential to preserve crestal bone level and prevent marginal soft tissue recession. According to a meta-analysis of 15 randomized-controlled trials, the estimated mean (SD) bone resorption for GBR in lateral ridge augmentation throughout the 6-month healing period was 1.22-0.28 mm. As a result, a 3.5 mm thickness of labial graft at all levels may be necessary following wound closure to compensate for potential graft loss.

Traditional bone augmentation is often dependent on the operator's skill, therefore virtually digital guided bone regeneration (GBR) process offers the digital options for precise and controllable bone augmentation in the field of oral implantology .

Specific aim: to compare the contour of bone augmentation (peri-implant bone volume) between various (GBR) procedures in patients with lateral alveolar ridge defect and simultaneous implantation.

Hypothesis: patients with lateral alveolar ridge defect and simultaneous implantation subjected to a 3D printing surgical template with GBR are associated with radiographic evidence of more labial graft thickness and volume stability after six months post-surgical than patients with conventional GBR protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients between the ages of 18 and 65 with edentulous ridge and seek for implant replacement.
2. In the anterior region, there is a labial bone defect.
3. Patients need the surgery in the first place to compensate for bone loss around implant.

Exclusion Criteria:

1. Systemic disorders that are out of control.
2. Heavy smokers (those who smoke more than 20 per day).
3. Women who are pregnant or nursing.
4. Thin gingival bio-type.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in Radiographic assessment for all patients underwent Cone beam computed tomography (CBCT) scans | baseline, immediately after and 6 months after surgery
  The postoperative CBCT DICOM images were converted to STL files and overlaid over the preoperative CBCT.The thickness of the labial bone graft was measured from the labial outline of the bone graft to the implant as a result of the procedure. (T0-T5) Perpendicular to the simulated implant in the bucco-oral cross-sectional picture. The distance (width in millimeter) between the implant and the labial contour of the graft, which indicated the thickness of the labial bone graft, was measured at the implant shoulder (T0), as well as at 1, 2, 3, 4, and 5 mm apical to the implant shoulder (T1-T5).
  For each site, the standard deviation of T0, T1, and T2 (SDC) was calculated, which represents the uniformity of the graft contour in the coronal area.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry-Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang M, Zhang X, Li Y, Mo A. The Influence of Different Guided Bone Regeneration Procedures on the Contour of Bone Graft after Wound Closure: A Retrospective Cohort Study. Materials (Basel). 2021 Jan 27;14(3):583. doi: 10.3390/ma14030583. PMID 33513735